CLINICAL TRIAL: NCT00377962
Title: Nordic Everolimus (Certican) Trial in Heart and Lung Transplantation: Results at 24 Months
Brief Title: Nordic Everolimus (Certican) Trial in Heart and Lung Transplantation
Acronym: NOCTET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRAD001AIC01
Record Dates: First submitted 2006-09-15; First posted 2006-09-19 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Disorder Related to Cardiac Transplantation
Keywords: thoracic transplant recipients; everolimus; immunosuppressants
MeSH Terms: interventions — Everolimus; Mycophenolic Acid; Calcineurin Inhibitors; Steroids

ARMS (2):
- Everolimus + CNI reduction (Experimental): Everolimus (3-8 ng/mL) + CNI reduction ± MPA/AZA ± steroids. Everolimus 0.75-1.5 mg twice daily. Dose adjusted to target blood concentration in the range 3-8 ng/mL. CNI reduction (reduced 50-70%): target of achieving a cyclosporine A (CsA) trough level < 75 ng/mL or a tacrolimus trough level < 4 ng/mL. MPA was reduced by 25%,upon CNI reduction. If participants were treated with AZA ( alternative to MPA) no dose reduction was needed. Steroid treatment was according to local practice.
  Interventions: Drug: Everolimus; Drug: Calcineurin inhibitors (CNI); Drug: Steroids
- Control (Active Comparator): CNI ± MPA/AZA ± steroids. In the standard CNI arm, all immunosuppressants including mycophenolic acid (MPA) and azathioprine (AZA) continued unchanged as per local practice. Steroid treatment was according to local practice.
  Interventions: Drug: Mycophenolic acid (MPA)/azathioprine (AZA); Drug: Calcineurin inhibitors (CNI); Drug: Steroids

INTERVENTIONS:
Drug: Everolimus — 0.75-1.5 mg twice daily. At the week 1 visit and thereafter, the dose was adjusted to target blood concentration in the range 3-8 ng/mL.
  Other Names: Certican
  Arms: Everolimus + CNI reduction
Drug: Mycophenolic acid (MPA)/azathioprine (AZA) — In the standard CNI arm, all immunosuppressants including (MPA) and azathioprine (AZA) continued unchanged as per local practice.
  Other Names: Neoral®/Prograf®
  Arms: Control
Drug: Calcineurin inhibitors (CNI) — Calcineurin inhibitors include cyclosporine, pimecrolimus, and tacrolimus.
Drug: Steroids — Steroid treatment was according to local practice. If steroids were given, the baseline dose of prednisone or equivalent was to be kept unchanged for all treatment groups for the total study duration, unless a medical condition dictated a change.

SUMMARY:
This study investigated whether initiation of everolimus together with reduction of calcineurin inhibitors (CNI) in maintenance heart or lung transplant patients with renal impairment would improve renal function.

ELIGIBILITY:
Inclusion criteria:

* Patients who have undergone a heart or lung transplantation more than 12 months ago.
* Patients receiving Neoral® or Prograf®.
* Patients with a measured or calculated glomerular filtration rate (GFR) > 20 and < 70 mL/min/1.73m^2. For patients with a GFR > 60 and < 70 mL/min/1.73m^2, a deteriorated renal function since the time of transplantation must be documented by at least one post-transplant GFR level that is > 10% above the GFR level at the time of inclusion.
* Patients willing and capable of giving written informed consent for study participation and able to participate in the study for 12 months.
* Females of potential childbearing age must have a negative serum pregnancy test within 7 days prior to enrollment. Effective contraception must be used during the trial and for 6 weeks following discontinuation of the study medication, even where there has been a history of infertility.

Exclusion criteria:

* Patients who are recipients of multiple organ transplants.
* Patients with measured GFR < 20 mL/min/1.73m^2 or > 70 mL/min/1.73m^2.
* Patients with a treated acute rejection episode within the last 3 months.
* Patients with a platelet count of < 50,000/mm^3 or with a white blood cell count of ≤ 2,500/mm^3 or with a hemoglobin value < 8 g/dL.
* Presence of severe hypercholesterolemia (≥ 8.0 mmol/L) or hypertriglyceridemia (≥ 6.0 mmol/L) despite conventional lipid lowering treatment.
* Patients currently treated or who have been treated with a mammalian target of rapamycin (mTOR) inhibitor.
* Patients who have received an investigational drug within 4 weeks.
* Patients who are human immunodeficiency virus positive or who have a current severe systemic infection requiring continued therapy according to investigator judgment.
* Present use of any immunosuppressive drugs other than Neoral®/Prograf®, mycophenolic acid/azathioprine (MPA/AZA), and/or steroids.
* Patients with a known hypersensitivity to drugs similar to everolimus.
* Symptoms of significant mental illness which, in the opinion of the investigator, may interfere with the patient's ability to comply with the protocol. History of drug or alcohol abuse within 1 year of baseline.
* Inability to cooperate or communicate with the investigator.
* Patients with any past (within the last 5 years) or present malignancy other than excised squamous or basal cell carcinoma.
* Females of childbearing potential that are planning to become pregnant, who are pregnant and/or lactating, or who are unwilling to use effective means of contraception.
* Patients with a planned coronary revascularization or patients who have experienced a major adverse cardiovascular event (MACE) within the last 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2005-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Denmark (2):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen
- Novartis Investigative Site, Oslo, Norway
- Sweden (3):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Norum HM, Michelsen AE, Lekva T, Arora S, Otterdal K, Olsen MB, Kong XY, Gude E, Andreassen AK, Solbu D, Karason K, Dellgren G, Gullestad L, Aukrust P, Ueland T. Circulating delta-like Notch ligand 1 is correlated with cardiac allograft vasculopathy and suppressed in heart transplant recipients on everolimus-based immunosuppression. Am J Transplant. 2019 Apr;19(4):1050-1060. doi: 10.1111/ajt.15141. Epub 2018 Nov 5. PMID 30312541
- [Derived] Arora S, Erikstad I, Ueland T, Sigurdardottir V, Ekmehag B, Jansson K, Eiskjaer H, Botker HE, Mortensen SA, Saunamaki K, Gude E, Ragnarsson A, Solbu D, Aukrust P, Gullestad L. Virtual histology assessment of cardiac allograft vasculopathy following introduction of everolimus--results of a multicenter trial. Am J Transplant. 2012 Oct;12(10):2700-9. doi: 10.1111/j.1600-6143.2012.04234.x. Epub 2012 Sep 7. PMID 22958738
- [Derived] Arora S, Gude E, Sigurdardottir V, Mortensen SA, Eiskjaer H, Riise G, Mared L, Bjortuft O, Ekmehag B, Jansson K, Simonsen S, Aukrust P, Solbu D, Iversen M, Gullestad L. Improvement in renal function after everolimus introduction and calcineurin inhibitor reduction in maintenance thoracic transplant recipients: the significance of baseline glomerular filtration rate. J Heart Lung Transplant. 2012 Mar;31(3):259-65. doi: 10.1016/j.healun.2011.12.010. PMID 22333403

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 12-month study in maintenance heart and lung transplant patients with a follow-up period of an additional 12 months. Results to 24 months are presented. Patients were randomized to continue their current calcineurin inhibitors (CNI) based regimen or to start everolimus with reduction of CNI blood levels.
Period: Core Study: 0-12 Months
Arm/Group | Everolimus + CNI Reduction | Control
Started | 140 | 142
Completed | 112 | 133
Not Completed | 28 | 9
Not completed — Adverse Event | 18 | 2
Not completed — Death | 3 | 0
Not completed — Withdrew Consent | 5 | 2
Not completed — Administrative Reason | 1 | 1
Not completed — Unspecified reasons | 1 | 4
Period: Extension Study: 12-24 Months
Arm/Group | Everolimus + CNI Reduction | Control
Started | 108 | 127
Completed | 98 | 123
Not Completed | 10 | 4
Not completed — Death | 1 | 1
Not completed — Adverse Event | 8 | 0
Not completed — Abnormal laboratory value | 1 | 0
Not completed — Unspecified reason | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus + CNI Reduction | Control | Total
Number analyzed (Participants) | 140 | 142 | 282
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (9.5) | 56.4 (10.7) | 57.8 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 40 | 77
  Male | 103 | 102 | 205

OUTCOME MEASURES:

1. Primary Outcome: Change in Measured Glomerular Filtration Rate (mGFR) From Baseline to Month 12
Description: Renal function was assessed by determining the measured glomerular filtration rate (mGFR) using creatinine ethylenediamine tetraacetic acid (Cr-EDTA) clearance or an equivalent method. A positive change score indicates improved renal function.
Time Frame: Baseline to Month 12
Population: Intent-to-treat (ITT) population: All randomized patients who were given at least 1 dose of study drug and had at least 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Everolimus + CNI Reduction | Control
Number analyzed (Participants) | 114 | 132
mL/min
  Baseline | 48.6 (15.1) | 48.0 (13.2)
  Month 12 | 53.2 (15.7) | 47.5 (16.1)
  Change from Baseline | 4.6 (10.4) | -0.5 (9.0)

2. Secondary Outcome: Change in Measured Glomerular Filtration Rate (mGFR) From Baseline to End of Study (Month 24)
Description: as for outcome 1
Time Frame: Baseline to end of study (Month 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Everolimus + CNI Reduction | Control
Number analyzed (Participants) | 103 | 119
mL/min
  Month 0 | 49.3 (14.7) | 49.1 (13.0)
  Month 24 | 52.5 (16.4) | 46.8 (15.2)
  Change | 3.2 (12.3) | -2.4 (9.0)

3. Secondary Outcome: Change in Serum Creatinine From Baseline to End of Study (Month 24)
Description: Renal function was assessed by determining serum creatinine using standard laboratory methods. A positive change score indicates improved renal function.
Time Frame: Baseline to end of study (Month 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Everolimus + CNI Reduction | Control
Number analyzed (Participants) | 114 | 132
μmol/L
  Month 0 | 126 (30) | 129 (29)
  Month 24 | 126 (64) | 132 (37)
  Change | 0 (53) | 3 (23)

4. Secondary Outcome: Number of Patients With Biopsy-proven Acute Rejection From Month 12 to End of Study (Month 24)
Description: Biopsy-proved acute rejection was defined as a treated acute rejection confirmed by biopsy, graded locally according to the International Society for Heart & Lung Transplantation (ISHLT) criteria. A treated acute rejection was defined as an acute rejection clinically suspected, whether biopsy-proven or not, which had been treated and confirmed by the investigator according to the response to therapy.
Time Frame: Month 12 to end of study (Month 24)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Everolimus + CNI Reduction | Control
Number analyzed (Participants) | 108 | 127
Participants | 6 | 5

5. Secondary Outcome: Number of Patients Who Died and Number of Patients With Graft Loss From Month 12 to End of Study (Month 24)
Description: Number of patients not alive and number of patients with loss of their graft.
Time Frame: Month 12 to end of study (Month 24)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Everolimus + CNI Reduction | Control
Number analyzed (Participants) | 108 | 127
Participants
  Death | 3 | 0
  Graft Loss | 0 | 0

6. Secondary Outcome: Number of Patients in Need of Dialysis From Month 12 to End of Study (Month 24)
Time Frame: Month 12 to end of study (Month 24)
Population: The intent-to-treat (ITT) population consisted of all patients as randomized, who were given at least one dose of study drug and had at least one post-baseline assessment. (Extension study)
Measure: Number; unit: Participants
Arm/Group | Everolimus + CNI Reduction | Control
Number analyzed (Participants) | 108 | 127
Participants | 0 | 2

7. Secondary Outcome: Change in Forced Expiratory Volume in 1 Second (FEV1) From Baseline to End of Study (Month 24) in the Lung Transplant Subgroup
Description: Forced expiratory volume in 1 second (FEV1) was measured by spirometry conducted according to internationally accepted standards. FEV1 is the volume delivered in the first second of a forced vital capacity (FVC) maneuver. A positive change score indicates improved lung function.
Time Frame: Baseline to end of study (Month 24)
Population: Patients in the lung transplant subgroup of the intent-to-treat (ITT) population which included all randomized patients who were given at least 1 dose of study drug and had at least 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Everolimus + CNI Reduction | Control
Number analyzed (Participants) | 36 | 40
Liters | -0.2 (0.2) | -0.1 (0.2)

8. Secondary Outcome: Change in Forced Vital Capacity (FVC) From Baseline to End of Study (Month 24) in the Lung Transplant Subgroup
Description: Forced vital capacity (FVC) was measured by spirometry conducted according to internationally accepted standards. FVC is the volume delivered during an expiration made as forcefully and completely as possible starting from full inspiration. A positive change score indicates improved lung function.
Time Frame: Baseline to end of study (Month 24)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Everolimus + CNI Reduction | Control
Number analyzed (Participants) | 36 | 40
Liters | -0.2 (0.3) | -0.1 (0.4)

9. Secondary Outcome: Change in Left Ventricular Function (Diameter and Thickness Parameters) From Baseline to End of Study (Month 24) in the Heart Transplant Subgroup
Description: Left ventricular function was assessed by echocardiography which was performed according to local routine practice. Echocardiography parameters were left ventricular end diastolic diameter (LVEDD), left ventricular end systolic diameter (LVESD), interventricular septal wall thickness (IVSTd), and posterior wall thickness (PWTd). A positive change score indicates improved left ventricular function.
Time Frame: Baseline to end of study (Month 24)
Population: Patients in the heart transplant subgroup of the intent-to-treat (ITT) population which included all randomized patients who were given at least 1 dose of study drug and had at least 1 post-baseline assessment.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Everolimus + CNI Reduction | Control
Number analyzed (Participants) | 56 | 73
cm
  LVEDD | -0.1 (0.8) | -0.0 (0.4)
  LVESD: number analyzed (Participants) | 42 | 57
  LVESD | 0.1 (0.7) | 0.1 (0.6)
  IVSTd: number analyzed (Participants) | 43 | 57
  IVSTd | -0.4 (2.4) | -0.1 (1.2)
  PWTd: number analyzed (Participants) | 43 | 56
  PWTd | -0.5 (2.1) | -0.1 (1.1)

10. Secondary Outcome: Change in Left Ventricular Function (Filling and Ejection Fraction Parameters) From Baseline to End of Study (Month 24) in the Heart Transplant Subgroup
Description: Left ventricular function was assessed by echocardiography which was performed according to local routine practice. Echocardiography parameters were filling fraction (FF) and ejection fraction (EF). A positive change score indicates improved left ventricular function.
Time Frame: Baseline to end of study (Month 24)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Everolimus + CNI Reduction | Control
Number analyzed (Participants) | 59 | 71
percentage
  EF | -0.6 (8.5) | 0.1 (7.9)
  FF: number analyzed (Participants) | 42 | 57
  FF | 0 (1) | 0 (1)

11. Secondary Outcome: Mean Days of Hospitalization From Baseline to End of Study (Month 24)
Time Frame: Baseline to end of study (Month 24)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Everolimus + CNI Reduction | Control
Number analyzed (Participants) | 108 | 127
Days | 8.5 (7.4) | 16.2 (19.3)

12. Secondary Outcome: Number of Patients Discontinued From the Study Due to Adverse Events From Month 12 to End of Study (Month 24)
Time Frame: Month 12 to end of study (Month 24)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Everolimus + CNI Reduction | Control
Number analyzed (Participants) | 108 | 127
Participants
  Total discontinued due to AE(s) | 8 | 0
  Pulmonary embolism | 2 | 0
  Skin problems | 1 | 0
  Hypercholesterolemia | 1 | 0
  Stroke | 1 | 0
  Muscular pain | 1 | 0
  Diarrhea | 1 | 0
  Edema | 1 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Safety population stratified by sub groups (heart patients and lung patients) and duration of core study and extension study.
Groups:
- Control: 12 Month Heart: Subgroup of "Control" group with heart patients at 12 months. CNI ± MPA/AZA ± steroids. In the standard CNI arm, all immunosuppressants including mycophenolic acid (MPA) and azathioprine (AZA) continued unchanged as per local practice. Steroid treatment was according to local practice.
- Everolimus + CNI Reduction: 12 Month Heart: Subgroup of "everolimus + CNI reduction" group with heart patients at 12 months. Everolimus (3-8 ng/mL) + CNI reduction ± MPA/AZA ± steroids. Everolimus 0.75-1.5 mg twice daily. Dose adjusted to target blood concentration in the range 3-8 ng/mL. CNI reduction (reduced 50-70%): target of achieving a cyclosporine A (CsA) trough level < 75 ng/mL or a tacrolimus trough level < 4 ng/mL. MPA was reduced by 25%, upon CNI reduction. If participants were treated with AZA ( alternative to MPA) no dose reduction was needed. Steroid treatment was according to local practice.
- Control: 12 Month Lung: Subgroup of "control" group with lung patients at 12 months. CNI ± MPA/AZA ± steroids. In the standard CNI arm, all immunosuppressants including mycophenolic acid (MPA) and azathioprine (AZA) continued unchanged as per local practice. Steroid treatment was according to local practice.
- Everolimus+CNI Reduction: 12 Month Lung: Subgroup of "everolimus + CNI reduction" group with lung patients at 12 months. Everolimus (3-8 ng/mL) + CNI reduction ± MPA/AZA ± steroids. Everolimus 0.75-1.5 mg twice daily. Dose adjusted to target blood concentration in the range 3-8 ng/mL. CNI reduction (reduced 50-70%): target of achieving a cyclosporine A (CsA) trough level < 75 ng/mL or a tacrolimus trough level < 4 ng/mL. MPA was reduced by 25%, upon CNI reduction. If participants were treated with AZA ( alternative to MPA) no dose reduction was needed. Steroid treatment was according to local practice.
- Control: 24 Month Heart: Subgroup of "Control" group with heart patients at 24 months. CNI ± MPA/AZA ± steroids. In the standard CNI arm, all immunosuppressants including mycophenolic acid (MPA) and azathioprine (AZA) continued unchanged as per local practice. Steroid treatment was according to local practice.
- Everolimus + CNI Reduction: 24 Month Heart: Subgroup of "everolimus + CNI reduction" group with heart patients at 24 months. Everolimus (3-8 ng/mL) + CNI reduction ± MPA/AZA ± steroids. Everolimus 0.75-1.5 mg twice daily. Dose adjusted to target blood concentration in the range 3-8 ng/mL. CNI reduction (reduced 50-70%): target of achieving a cyclosporine A (CsA) trough level < 75 ng/mL or a tacrolimus trough level < 4 ng/mL. MPA was reduced by 25%, upon CNI reduction. If participants were treated with AZA ( alternative to MPA) no dose reduction was needed. Steroid treatment was according to local practice.
- Control: 24 Month Lung: Subgroup of "Control" group with lung patients at 24 months. CNI ± MPA/AZA ± steroids. In the standard CNI arm, all immunosuppressants including mycophenolic acid (MPA) and azathioprine (AZA) continued unchanged as per local practice. Steroid treatment was according to local practice.
- Everolimus + CNI Reduction: 24 Month Lung: Subgroup of "everolimus + CNI reduction" group with lung patients at 24 months. Everolimus (3-8 ng/mL) + CNI reduction ± MPA/AZA ± steroids. Everolimus 0.75-1.5 mg twice daily. Dose adjusted to target blood concentration in the range 3-8 ng/mL. CNI reduction (reduced 50-70%): target of achieving a cyclosporine A (CsA) trough level < 75 ng/mL or a tacrolimus trough level < 4 ng/mL. MPA was reduced by 25%, upon CNI reduction. If participants were treated with AZA ( alternative to MPA) no dose reduction was needed. Steroid treatment was according to local practice.
Arm/Group | Control: 12 Month Heart | Everolimus + CNI Reduction: 12 Month Heart | Control: 12 Month Lung | Everolimus+CNI Reduction: 12 Month Lung | Control: 24 Month Heart | Everolimus + CNI Reduction: 24 Month Heart | Control: 24 Month Lung | Everolimus + CNI Reduction: 24 Month Lung
Serious Adverse Events (participants affected / at risk) | 23/96 | 40/94 | 17/46 | 25/46 | 31/86 | 25/69 | 21/41 | 16/39
Other Adverse Events (participants affected / at risk) | 48/96 | 75/94 | 33/46 | 42/46 | 33/86 | 29/69 | 21/41 | 27/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control: 12 Month Heart (N=96) | Everolimus + CNI Reduction: 12 Month Heart (N=94) | Control: 12 Month Lung (N=46) | Everolimus+CNI Reduction: 12 Month Lung (N=46) | Control: 24 Month Heart (N=86) | Everolimus + CNI Reduction: 24 Month Heart (N=69) | Control: 24 Month Lung (N=41) | Everolimus + CNI Reduction: 24 Month Lung (N=39)
Anaemia NOS (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure NOS (Cardiac disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Coronary artery atheroma haemorrhage (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease NOS (Cardiac disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Oedema NOS (Cardiac disorders) | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0
Pulmonary oedema NOS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Right ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain NOS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Appendicitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea NOS (Gastrointestinal disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 0
Diverticulitis NOS (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Food poisoning NOS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia NOS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis NOS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal disorder NOS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting NOS (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Compartment syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhage NOS (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain NOS (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Graft rejection (Immune system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Heart transplant rejection (Immune system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity NOS (Immune system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Brain abscess NOS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis NOS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis acute NOS (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Cholecystitis acute NOS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis NOS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection NOS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Epididymitis NOS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gastroenteritis NOS (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1
Infection NOS (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Lobar pneumonia NOS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection NOS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia NOS (Infections and infestations) | 3 | 7 | 3 | 6 | 2 | 0 | 7 | 5
Pneumonia aspergilla (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pseudomonas aeruginosa infection NOS (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pyelonephritis NOS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis NOS (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis NOS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection NOS (Infections and infestations) | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Urinary tract infection NOS (Infections and infestations) | 1 | 3 | 1 | 0 | 1 | 2 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fracture NOS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Leg fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arteriogram coronary (Investigations) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Biopsy lung (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung function abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung function decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte morphology NOS abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pericardial drainage (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition NOS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthritis NOS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intervertebral disc prolapse (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sciatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Benign adrenal neoplasm NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer female NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Carcinoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung cancer stage unspecified (exc metas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Malignant melanoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Prostate cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Skin carcinoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 1 | 1 | 0 | 0 | 1 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Burning sensation NOS (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident NOS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (exc vertigo) (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy NOS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine NOS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Monoparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Restless leg syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Syncope aggravated (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nephropathy NOS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure NOS (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Renal impairment NOS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma NOS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 1 | 2 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Excessive bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mediastinal emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 6 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Respiratory failure (exc neonatal) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis NOS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic foot ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angioplasty (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial lesion excision (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hip arthroplasty (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Leg amputation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Operation NOS (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Suture removal (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arterial stenosis NOS (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cerebral artery thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension aggravated (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intracranial haemorrhage NOS (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis NOS (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Postural hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Vascular disorders) | 1 | 1 | 2 | 2 | 1 | 2 | 1 | 1
Pulmonary hypertension NOS (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Subarachnoid haemorrhage NOS (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Vascular disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Venous thrombosis NOS (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Venous thrombosis deep limb (Vascular disorders) | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control: 12 Month Heart (N=96) | Everolimus + CNI Reduction: 12 Month Heart (N=94) | Control: 12 Month Lung (N=46) | Everolimus+CNI Reduction: 12 Month Lung (N=46) | Control: 24 Month Heart (N=86) | Everolimus + CNI Reduction: 24 Month Heart (N=69) | Control: 24 Month Lung (N=41) | Everolimus + CNI Reduction: 24 Month Lung (N=39)
Leucopenia NOS (Blood and lymphatic system disorders) | 0 | 8 | 0 | 8 | 1 | 1 | 0 | 1
Oedema NOS (Cardiac disorders) | 10 | 24 | 3 | 14 | 9 | 4 | 2 | 5
Epidermal naevus (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 1 | 0 | 3 | 0
Diarrhoea NOS (Gastrointestinal disorders) | 4 | 15 | 3 | 7 | 0 | 4 | 1 | 3
Gastritis NOS (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 5 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 1 | 2 | 2 | 1 | 1 | 2
Fall (General disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 5 | 6 | 2 | 2 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 6 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Bronchitis NOS (Infections and infestations) | 0 | 5 | 3 | 2 | 0 | 0 | 2 | 2
Infection NOS (Infections and infestations) | 0 | 3 | 1 | 0 | 3 | 2 | 2 | 2
Influenza (Infections and infestations) | 5 | 2 | 2 | 1 | 1 | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 15 | 18 | 12 | 11 | 12 | 7 | 7 | 8
Pneumonia NOS (Infections and infestations) | 5 | 3 | 2 | 5 | 1 | 0 | 0 | 3
Upper respiratory tract infection NOS (Infections and infestations) | 1 | 2 | 6 | 9 | 2 | 2 | 4 | 6
Urinary tract infection NOS (Infections and infestations) | 0 | 3 | 3 | 4 | 1 | 1 | 2 | 3
Blood creatinine increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 | 0 | 3 | 6 | 1 | 2 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 4 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 2 | 3 | 0 | 1 | 1 | 1
Arthritis NOS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 7 | 1 | 1 | 2 | 0 | 0 | 0
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0 | 1 | 2 | 1 | 0 | 0
Headache NOS (Nervous system disorders) | 7 | 7 | 3 | 5 | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 3 | 3 | 0 | 3 | 1 | 1
Excessive bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Acne NOS (Skin and subcutaneous tissue disorders) | 0 | 11 | 0 | 1 | 0 | 0 | 0 | 1
Hypertension NOS (Vascular disorders) | 5 | 4 | 4 | 6 | 0 | 3 | 2 | 3
Hypertension aggravated (Vascular disorders) | 0 | 5 | 1 | 1 | 3 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.